CLINICAL TRIAL: NCT02669966
Title: Live Kidney Donors With Positive Anti-HCV Antibody, But Negative HCV PCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201500543
Record Dates: First submitted 2016-01-27; First posted 2016-02-01 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: ESRD; Hepatitis C
Keywords: Kidney Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic; Hepatitis C | interventions — Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Donor candidates with their intended recipients who meet criteria will be enrolled into this, the sole arm of our study. Donor-recipient pairs will be screened to meet criteria, and will proceed to kidney transplantation and post-transplant monitoring
  Interventions: Procedure: Kidney transplantation

INTERVENTIONS:
Procedure: Kidney transplantation — Once the donor and recipient candidates have met inclusion criteria and cleared study-specific as well as standard of care screening, they will proceed to live-donor kidney transplantation and subsequent post-transplant monitoring

SUMMARY:
It is well recognized that a subset of patients who contracts Hepatitis C virus (HCV) spontaneously clears the virus. Such individuals are anti-HCV antibody positive, yet HCV RNA PCR negative in the blood. While they have not been considered candidates for live kidney donation in the past, with the recent availability of novel anti-HCV drugs with >95% cure rates, they now represent a potential pool of donor candidates, especially since the risk for transmission of HCV to the recipient is extremely low. The investigators goal is to demonstrate that live kidney donation from anti-HCV positive, HCV RNA PCR negative individuals is safe and carries a negligible risk of viral transmission to the recipient.

DETAILED DESCRIPTION:
Individuals who test positive for anti-HCV IgG antibody, but who have negative blood HCV RNA PCR are generally considered to have been infected with HCV but to have cleared the the virus spontaneously. However, due to the general conservative approach of living donor kidney transplant programs, these individuals are not considered potential live kidney donors, despite being considered at extremely low risk for HCV transmission to the recipient. This reluctance stems from past experiences with post-transplant HCV complications, both hepatic (e.g. cirrhosis) and extra-hepatic (e.g. transplant glomerulonephritis) and from the fact that the historical mainstay of HCV treatment, interferon, was poorly tolerated, had low cure rates, and caused transplant rejection. Now, however, highly effective novel therapeutics may transform the way transplant physicians and patients think about HCV-positive donated kidneys.

With these new agents, the current cure rates for HCV now exceed 95%. A recent report demonstrated high cure rates even in the liver transplant setting, suggesting that immunosuppression does not impede eradication and that interactions between HCV and transplant drugs can be successfully managed. Thus, while the risk of transmission of infection from anti-HCV antibody positive, HCV PCR-negative is not known, if transmission were to occur, treatment is now possible, to the point where transplant professionals are beginning to advocate using anti-HCV Ab positive individuals as donors for HCV-negative recipients. A group in Barcelona reported transplantation of a live donor kidney from a donor treated with an anti-HCV regimen that achieved a sustained virological response to her spouse with no transmission of infection.

The main area of concern seems to be what is described as "occult HCV infection"- the presence of HCV RNA in peripheral blood mononuclear cells and organ tissue by ultrasensitive assays in the absence of detectable RNA in the serum. However, this entity is itself controversial, and its significance is uncertain, with inadequately described risk of transmission. If HCV were transmitted and successfully treated, another concern is the potential residual risks of viral complications, even though these have not been evident in any previous trials. Finally, a major concern is financial, as HCV treatment currently costs more than $80,000 for a 3-month regimen. However, chronic hemodialysis costs upwards of $100,000 per year when all costs are considered, while kidney transplantation costs only about $20,000 per year after the first year. Thus, over time, even after treatment for CMV infection, if it is required, kidney transplantation would result in an overall cost savings to the health care system.

Given the unknown, though generally considered very low risk of transmission of HCV from an antibody-positive, PCR-negative individual, combined with the wide availability of effective treatment for HCV infection, it is felt that the recipient is not exposed to a high risk of infection in such a transplant. Furthermore, this small risk needs to be weighed against the risk of staying on dialysis, which carries a mortality rate of 6.5-7.4 times that of the general population and 4.6-5.9 times that of the renal transplant population. The case becomes even more compelling when considering patients with a high risk of deterioration if they continue dialysis (elderly, diabetics, and those with cardiovascular disease), disadvantageous blood types, and those with broad sensitization, with extremely limited compatible donor options. Given the proven survival benefit of kidney transplantation in patients with chronic HCV, there is ample reason to believe that providing HCV positive kidneys and HCV therapy (if indeed required) to HCV negative recipients will lead to better outcomes than those associated with remaining on dialysis.

ELIGIBILITY:
Inclusion Criteria:

Donor inclusion criteria:

* The donor candidate must be anti-HCV positive by ELISA and HCV RNA negative by PCR, with both tests repeated for confirmation, as per standard protocol.
* The donor must be evaluated and cleared by Hepatology, which is currently the standard of care for HCV seropositive individuals.
* The donor must meet criteria for living kidney donation and be approved by the UF Health Shands Kidney Transplant Medical Review Board.

Recipient inclusion criteria:

* The recipient may be HCV antibody negative or anti-HCV antibody positive but HCV RNA negative by PCR.
* The recipient must meet the criteria for kidney transplantation and be approved by the UF Health Kidney Transplant Program Medical Review Board.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-03; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Maintenance of HCV seronegativity | 3 months
  At 3 months post-transplant, recipients will be screened for HCV seropositivity. A negative seropositive result will conclude the recipient's participation in the study

CONTACTS AND LOCATIONS:
Overall Officials: Karl Womer, MD, Principal Investigator — Univesity of Florida
Locations (1):
- Shands at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afdhal N, Zeuzem S, Kwo P, Chojkier M, Gitlin N, Puoti M, Romero-Gomez M, Zarski JP, Agarwal K, Buggisch P, Foster GR, Brau N, Buti M, Jacobson IM, Subramanian GM, Ding X, Mo H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Mangia A, Marcellin P; ION-1 Investigators. Ledipasvir and sofosbuvir for untreated HCV genotype 1 infection. N Engl J Med. 2014 May 15;370(20):1889-98. doi: 10.1056/NEJMoa1402454. Epub 2014 Apr 11. PMID 24725239
- [Background] Schold J, Srinivas TR, Sehgal AR, Meier-Kriesche HU. Half of kidney transplant candidates who are older than 60 years now placed on the waiting list will die before receiving a deceased-donor transplant. Clin J Am Soc Nephrol. 2009 Jul;4(7):1239-45. doi: 10.2215/CJN.01280209. Epub 2009 Jun 18. PMID 19541814
- [Background] Cruzado JM, Gil-Vernet S, Castellote J, Bestard O, Melilli E, Grinyo JM. Successful treatment of chronic HCV infection should not preclude kidney donation to an HCV negative recipient. Am J Transplant. 2013 Oct;13(10):2773-4. doi: 10.1111/ajt.12400. Epub 2013 Aug 6. No abstract available. PMID 23919533
- [Background] Baid-Agrawal S, Schindler R, Reinke P, Staedtler A, Rimpler S, Malik B, Frei U, Berg T. Prevalence of occult hepatitis C infection in chronic hemodialysis and kidney transplant patients. J Hepatol. 2014 May;60(5):928-33. doi: 10.1016/j.jhep.2014.01.012. Epub 2014 Jan 18. PMID 24447875
- [Background] Halfon P, Martinot-Peignoux M, Cacoub P. The myth of occult hepatitis C infection. Hepatology. 2009 Nov;50(5):1675. doi: 10.1002/hep.23113. No abstract available. PMID 19585649
- [Background] Reddy KR EG, Flamm SL, et al. Ledipasvir/sofosbuvir with ribavirin for the treatment of HCV in patients with post-transplant recurrence: preliminary results of a prospective, multicenter study. Hepatology. 2014;60:200A.